CLINICAL TRIAL: NCT03908203
Title: Minimally Invasive Surgery Techniques for One-level Degenerative Lumbar Deformities Correction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The Study will be conducted in another research center. The Sponsor has changed.
Sponsor: Novosibirsk Research Institute of Traumatology and Orthopaedics n.a. Ya.L. Tsivyan (Other Government)
Collaborators: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NS02-02
Record Dates: First submitted 2019-04-06; First posted 2019-04-09 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-02

CONDITIONS: Intervertebral Disc Degeneration; Spinal Fusion
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Other)
  Interventions: Procedure: Minimally invasive one-level lumbar deformity correction

INTERVENTIONS:
Procedure: Minimally invasive one-level lumbar deformity correction — The study treatment represents modified technique of MIS TLIF: one level screws fixation using Wiltse approach at one side, the other side - percutaneously, one level decompression, correction of segmental deformity by performing vertebrotomy and then intervertebral fusion.

SUMMARY:
This study will be conducted at Research Institute of Traumatology and Orthopedics (NRITO) n.a. Ya.L.Tsivyan, Novosibirsk, Russia.

The current study is prospective pilot clinical study to demonstrate the possibility and effectiveness of performing modified technique of MIS TLIF, supplemented by segmental vertebrotomy, to correct segmental deformity of lumbar spine.

It is expected to enroll 10 patients aged 18-70 with segmental deformity of lumbar spine, caused by degenerative spondylolisthesis and/or degenerative stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Given written Informed Consent;
* Single-level segmental deformity caused by degenerative spondylolisthesis and/or degenerative stenosis at the one level of lumbar spine L4-L5 or L5-S1;
* Mono- and/or polyradicular leg pain and/or neurogenic claudication with or without back pain;
* Symptoms persisting for at least three months prior to surgery;
* Able and agree to fully comply with the clinical protocol and willing to adhere to follow-up schedule and requirements.

Exclusion Criteria:

* Lumbar deformation of non-degenerative etiology;
* Spondylolisthesis grade II or higher (25% slip or greater) of any etiology;
* Patient that has already undergone a lumbar fusion surgery;
* Other non-degenerative spinal conditions (e.g. infectious, traumatic, metabolic, inflammatory, neoplastic, structural or other pathology) that may have an impact on subject safety, wellbeing or the intent and conduct of the study
* Concurrent participation in another clinical study that may confound study results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Angle change at lumbar spine segment | At 1 Day of hospital discharge or 14th day of hospital stay (depends on what event comes first)
  Angle between endplates at the treated level of lumbar spine

SECONDARY OUTCOMES:
Improvement of Visual analog scale (VAS) back pain intensity | 3, 6, 12 months
  To observe the improvement of VAS back pain as compared to baseline through follow-up terms.
  Visual Analogue Scale (VAS) - patient-reported pain intensity (0 - no pain, 10 - unbearable pain).
Improvement of Visual analog scale (VAS) leg pain intensity | 3, 6, 12 months
  To observe the improvement of VAS leg pain as compared to baseline through follow-up terms.
  Visual Analogue Scale (VAS) - patient-reported pain intensity (0 - no pain, 10 - unbearable pain).
Improvement of Oswestry Disability Index (ODI) | 3, 6, 12 months
  To observe the improvement of ODI as compared to baseline through follow-up terms Oswestry Disability Index - patient-reported physical and household activity. Minimum - 0 % (the best result, the patient has no limitations in physical activity). Maximum - 100% (the worst result, patient is not physically active at all).
Fusion rate success | 12 months
  To observe the Fusion rate (I, II, III or IV grade according to Tan).
  Grade I - complete fusion; Grade II - partial fusion; Grade III - unipolar pseudarthrosis; Grade IV - bipolar pseudarthrosis.
Range of Motion | At 1 Day of hospital discharge or 14th day of hospital stay depends on what event comes first, 12 months
  To observe the disc mobility at the treated level
Sagittal balance parameters | At 1 Day of hospital discharge or 14th day of hospital stay depends on what event comes first, 12 months
  To observe sagittal balance as compared to baseline
Disc height | At 1 Day of hospital discharge or 14th day of hospital stay depends on what event comes first, 12 months
  To observe disc height at the treated level as compared to baseline
Blood loss | Day of surgery
  Blood loss
Surgery duration | Day of surgery
  Surgery duration

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandr V Krutko, PhD, MD, Principal Investigator — Novosibirsk Research Institute of Traumatology and Orthopaedics n.a. Ya.L. Tsivyan
Locations (1):
- Novosibirsk Research Institute of Traumatology and Orthopaedics n.a. Ya.L. Tsivyan, Novosibirsk, Russia